CLINICAL TRIAL: NCT00565838
Title: Clinical and Quality-of-Life Outcomes After Autologous Fascial Sling and Tension-Free Vaginal Tape: a Prospective Randomized Trial
Brief Title: Quality-of-Life Outcomes After Autologous Fascial Sling and TVT: a Prospective Randomized Trial
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: João Luiz Amaro/ Associate Professor, International Continence Society
Other Study IDs: upeclin/HC/FMB-Unesp-05
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Stress Urinary Incontinence
Keywords: Randomized study; surgical treatment; autologous fascial sling; TVT; stress urinary incontinence.
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2: G1 - Autologous Fascial Sling G2 - TVT
  Interventions: Procedure: AFS and TVT

INTERVENTIONS:
Procedure: AFS and TVT — Autologous Fascial Sling and Tension- Free Vaginal Tape
  Other Names: AFS; TVT

SUMMARY:
The objective of the study was to evaluate the impact AFS and TVT procedures on quality-of-life in incontinent women.

DETAILED DESCRIPTION:
Between January 2001 to March 2002, 41 women with a principal complaint of stress urinary incontinence were studied in a prospective trial. Based on results of no numerical variables (including patient's perception of improvement and satisfaction with treatment), the statistical test demonstrated the need for equal sized groups for the comparison. So, the total size of sample groups was previously established as at least 40 women.

These patients were randomly distributed, in a single-blind study, into two groups. Group G1 (n=21) was submitted to AFS and Group G2 (n=20) to TVT implant. Average age in G1 was 49 years (range 26-69), and in G2, 52 years (range 26-79). This study was approved by the Bioethics Commission of the School of Medicine - UNESP, Botucatu.

All the women underwent preoperative urodynamic study, using a Dynograph R.611 recorder, which confirmed stress urinary incontinence in all of them. Patients with involuntary detrusor contractions or preexisting bladder outlet obstruction (BOO) during urodynamic study were excluded of the study.

The clinical follow up and a subjective success rate was performed at 1, 6, and 12 months and then annually after hospital discharge. A questionnaire was used to obtain personal data, obstetric, gynecologic, family history, and subjective analysis of urine loss. Cure was defined as complete dryness with no usage of pads.

De novo urgency was considered when patients had no problem with urgency symptoms preoperatively presented these complaints after surgery persisting more than 1 month. These symptoms were based on clinical evaluation.

Long-term patients' satisfaction and impact on QoL were performed at 36 months after surgery. To evaluate the QoL a validated questionnaire (11) (King's Health Questionnaire) was used. Follow up range from 36 to 54 months (median: 44 months).

Body mass index (BMI) was calculated and classified according to Garrow. All patients underwent physical examination including stress test. The degree of pelvic organ prolapse was assessed and graded according to Baden et al.

Basal laboratory investigations (serum creatinine, complete blood count, chemical and microscopic urinalysis, urine culture) were all routinely performed. In exceptional cases (lithiasis history, urinary infection ) renal ultrasound and plain x-ray of the kidney, ureters and bladder were carried out.

In the immediate postoperative, endovenous tramadol (10 mg/mL-1) was used in patient controlled analgesia (PCA) pump. After an i.v. loading dose of 0.07 mL/Kg-1 (administered over a period of 30 min).

The Physiotherapy Service at each surgical procedure was responsible for carrying out the random assignment of patients in accordance with the casualty.

ELIGIBILITY:
Inclusion Criteria:

* Stress Urinary Incontinence

Exclusion Criteria:

* Detrusor obstruction or hyperactivity

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2001-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary outcome | Observational

CONTACTS AND LOCATIONS:
Overall Officials: João L Amaro, PhD MD, Principal Investigator — Department of Urology - UNESP
Locations (1):
- Medical School of Medicine, Botucatu, São Paulo, Brazil